CLINICAL TRIAL: NCT05583435
Title: Decreasing Physician Burnout With Professional Coaching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Joshua N. Khalili, MD, Assistant Clinical Professor of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-001542
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Burnout, Professional
Keywords: physician burnout; coaching; work engagement
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- One-on-one professional coaching (Experimental): One-on-one professional coaching (N=30). Six one-on-one coaching sessions via Zoom with one of two private professional coaches every other week for 3-4 months.
  The professional coaching method includes (but will not be limited to) the following themes: optimizing meaning and engagement in work, building social support and community, improving work efficiency, addressing workload and boundary setting, enhancing communication, and building leadership skills, pursuing hobbies and creation/innovation, and promoting self-compassion and self-care (with a focus on physical and mental health).
  Coach-guided activities/behavioral interventions are included with coaching sessions. These activities are reviewed with participants throughout the 3-4 month period and include, but are not limited to: Wheel of Life, visioning exercise, one page miracle: core values, purpose, and goals, buckets and mental models.
  Interventions: Behavioral: One-on-one professional coaching
- Small-group professional coaching with coach-guided activities/behavioral internventions (Experimental): Coach-facilitated small group professional coaching sessions and coach-guided activities/behavioral interventions (N=30). Six small-group coaching sessions via Zoom with one of two private professional coaches and three physician participants in each group, every other week for 3-4 months.
  The professional coaching method is similar to those receiving 1:1 professional coaching. The primary difference in this intervention group is that coaching sessions will be group-based with 3 physician participants.
  Interventions: Behavioral: Small-group professional coaching
- Delayed-entry group (placebo then one-on-one professional coaching) (Experimental): Delayed-Entry Group 3 (N=30). No intervention during the 90 day study period. Note: once participation in the pilot study has been completed for Groups 1 and 2, physicians participating in Group 3 will be offered to participate in six one-on-one sessions with a private professional coach over a 3 month period.
  The professional coaching method includes (but will not be limited to) the following themes: optimizing meaning and engagement in work, building social support and community, improving work efficiency, addressing workload and boundary setting, enhancing communication, and building leadership skills, pursuing hobbies and creation/innovation, and promoting self-compassion and self-care (with a focus on physical and mental health).
  Interventions: Behavioral: One-on-one professional coaching

INTERVENTIONS:
Behavioral: One-on-one professional coaching — One-on-one professional coaching
  Arms: Delayed-entry group (placebo then one-on-one professional coaching); One-on-one professional coaching
Behavioral: Small-group professional coaching — Small-group professional coaching
  Arms: Small-group professional coaching with coach-guided activities/behavioral internventions

SUMMARY:
The goal of this randomized control trial is to learn if professional coaching can help reduce physician burnout among physicians at UCLA. The main aims of the study are:

* To reduce burnout among physicians with professional coaching
* Improve work satisfaction and engagement, sense of self-efficacy and social support with professional coaching
* Determine the efficacy of one-on-one professional coaching and small group professional coaching combined with behavioral interventions/activities in reducing physician burnout and comparing these groups to one another and to a delayed-entry (control) group

Participants will be randomly assigned into one of three groups:

* Intervention Group 1: One-on-one coaching (N=30). Six one-on-one coaching sessions via Zoom with one of two private professional coaches every other week for 3-4 months.
* Intervention Group 2: Coach-facilitated group sessions and coach-guided activities/behavioral interventions (N=30). Six small-group coaching sessions via Zoom with one of two private professional coaches and three physician participants in each group, every other week for 3-4 months.
* Delayed-Entry Group 3 (N=30): No intervention during duration of study period. Note: once participation in the pilot study has been completed for Groups 1 and 2, physicians participating in Group 3 will be offered to participate in six one-on-one sessions with a private professional coach over a 3-4 month period.

Participants will complete several surveys that assess for burnout, work engagement and satisfaction, sense of social support and isolation, and areas of worklife) before the start, upon completion of the intervention and again at 6 months upon completion of the sessions for the delayed-entry group.

Each group also received coach-guided activities/behavioral interventions during coaching sessions. These activities will be sent by coaches to participates throughout the 3 month period and include, but are not limited to: Wheel of Life, visioning exercise, one page miracle: core values, purpose, and goals, buckets and mental models.

ELIGIBILITY:
Inclusion Criteria:

* Actively practicing UCLA department of medicine physicians who had at least two years of employment at UCLA

Exclusion Criteria:

* Current or anticipated (in the next 6 months) participation in one-on-one or group coaching provided by a professional coach

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2024-04-13 (Actual); Study Completion 2024-04-13 (Actual)

PRIMARY OUTCOMES:
Burnout | 90 days
  Physician burnout (as measured by emotional exhaustion, depersonalization and personal accomplishment) evaluated with the Maslach Inventory Scale

SECONDARY OUTCOMES:
Areas of Worklife | 90 days
  Workload, control, reward, community, fairness and values as measured by the Areas of Worklife Survey
Self-efficacy | 90 days
  Sense of self-efficacy as measured by New General Self-Efficacy Scale
Work Engagmement and Satisfaction | 90 days
  Measured by the Utrecht Work Engagement Scale
Social Support | 90 days
  Sense of social support and isolation as measured by the PROMIS Social Isolation Subscale and Social Provisions Scale

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Khalili, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maslach C, Jackson SE, Leiter MP. Maslach Burnout Inventory. 4th ed. Menlo Park, CA: Mind Garden; 2016
- [Background] Leiter MP, Maslach C. Six areas of worklife: a model of the organizational context of burnout. J Health Hum Serv Adm. 1999 Spring;21(4):472-89. PMID 10621016
- [Background] New General Self Efficacy Scale: Chen, G., Gully, S. M., & Eden, D. (2001). Validation of a new general self-efficacy scale. Organizational research methods, 4(1), 62-83
- [Background] Utrecht Work Engagement Scale: Schaufeli W, Bakker A. UWES: Utrecht Work Engagement Scale: preliminary manual [version 1.1, December 2004]. https://www.wilmarschaufeli.nl/publications/Schaufeli/Test%20Manuals/Test_manual_UWES_English.pdf.
- [Background] Hahn EA, DeWalt DA, Bode RK, Garcia SF, DeVellis RF, Correia H, Cella D; PROMIS Cooperative Group. New English and Spanish social health measures will facilitate evaluating health determinants. Health Psychol. 2014 May;33(5):490-9. doi: 10.1037/hea0000055. Epub 2014 Jan 20. PMID 24447188
- [Background] Social Provisions Scale: Cutrona CE, Russell DW. The provisions of social relationships and adaptation to stress. Advances in Personal Relationships. 1987;1:37-67.
- [Background] Dyrbye LN, Varkey P, Boone SL, Satele DV, Sloan JA, Shanafelt TD. Physician satisfaction and burnout at different career stages. Mayo Clin Proc. 2013 Dec;88(12):1358-67. doi: 10.1016/j.mayocp.2013.07.016. PMID 24290109
- [Background] Han S, Shanafelt TD, Sinsky CA, Awad KM, Dyrbye LN, Fiscus LC, Trockel M, Goh J. Estimating the Attributable Cost of Physician Burnout in the United States. Ann Intern Med. 2019 Jun 4;170(11):784-790. doi: 10.7326/M18-1422. Epub 2019 May 28. PMID 31132791
- [Background] Panagioti M, Panagopoulou E, Bower P, Lewith G, Kontopantelis E, Chew-Graham C, Dawson S, van Marwijk H, Geraghty K, Esmail A. Controlled Interventions to Reduce Burnout in Physicians: A Systematic Review and Meta-analysis. JAMA Intern Med. 2017 Feb 1;177(2):195-205. doi: 10.1001/jamainternmed.2016.7674. PMID 27918798
- [Background] Dyrbye LN, Shanafelt TD, Gill PR, Satele DV, West CP. Effect of a Professional Coaching Intervention on the Well-being and Distress of Physicians: A Pilot Randomized Clinical Trial. JAMA Intern Med. 2019 Oct 1;179(10):1406-1414. doi: 10.1001/jamainternmed.2019.2425. PMID 31380892
- [Derived] Khalili J, Miotto K, Wang T, Mafi JN, Kyababchyan E, Sanford J, Elashoff D, Brook J, Adebambo Y, Smith PI, Nguyen E, Yoo SM. Professional Coaching to Reduce Physician Burnout: A Randomized Clinical Trial. J Gen Intern Med. 2025 Jul 11. doi: 10.1007/s11606-025-09653-w. Online ahead of print. PMID 40643743